CLINICAL TRIAL: NCT02886585
Title: Phase II Trial of Pembrolizumab in Central Nervous System Metastases From Multiple Histologies
Brief Title: Pembrolizumab In Central Nervous System Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Priscilla Brastianos, Principal Investigator/ Physician, Cancer Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-153
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Brain Metastases
Keywords: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Previously Untreated Brain Metastases-Cohort A (Experimental): - Previously Untreated Brain Metastases
  * Baseline Brain MRI and PET CT
  * For all cohorts, pembrolizumab will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle. Treatment will be administered on an outpatient basis.
  * Brain MRI and PET/CT
  Interventions: Drug: Pembrolizumab; Radiation: MRI; Radiation: PET/CT
- Progressive Brain Metastases-Cohort B (Experimental): - Progressive Brain Metastases
  * Baseline Brain MRI and PET CT
  * For all cohorts, pembrolizumab will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle. Treatment will be administered on an outpatient basis.
  * Brain MRI and PET/CT
  Interventions: Drug: Pembrolizumab; Radiation: MRI; Radiation: PET/CT
- Neoplastic Meningitis-Cohort C (Experimental): * Neoplastic Meningitis
  * Histologically confirmed solid malignancy
  * Positive Cytology
    * Baseline Brain MRI
    * For all cohorts, pembrolizumab will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle. Treatment will be administered on an outpatient basis.
    * Brain MRI and PET/CT
  Interventions: Drug: Pembrolizumab; Radiation: MRI; Radiation: PET/CT
- 1-4 Brain Metastases from Melanoma Cohort D (Experimental): * 1-4 Brain Metastases from Melanoma
  * Clinical indication for stereostatic radiosurgery
  * Evaluable extracranial focus
    * For all cohorts, pembrolizumab will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle. In Cohort D, cycle 1 and 2 of pembrolizumab will be administered 3 weeks apart and stereotactic radiosurgery will be administered between cycles. Treatment will be administered on an outpatient basis.
    * Brain MRI and PET CT
  Interventions: Drug: Pembrolizumab; Radiation: MRI; Radiation: PET/CT; Procedure: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Pembrolizumab
Radiation: MRI
Radiation: PET/CT
Procedure: Stereotactic Radiosurgery
  Arms: 1-4 Brain Metastases from Melanoma Cohort D

SUMMARY:
This research study is studying Pembrolizumab as a possible treatment for this diagnosis for metastases in the central nervous system (brain and spinal cord).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

Pembrolizumab may help the immune system fight cancer.

The FDA (the U.S. Food and Drug Administration) has approved pembrolizumab FDA for some diseases that are being treated on this study, but not for central nervous system metastases. Researchers hope to study the effects of pembrolizumab. Many cancers use specific pathways (such as PD-1/PD-L1 and CTLA-4) to evade the body's immune system. Pembrolizumab works by blocking the PD-1/PD-L1 pathways and thus releasing the brakes on the immune system so it can stop or slow cancer.

Researchers hope to study the effects of pembrolizumab in cancer that has metastasized to the brain. These drugs work by stimulating the immune system to fight cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed disease from any solid tumor
* Participants must have measurable disease in the CNS, defined as at least one lesion that can be accurately measured in at least one dimension as ≥5 mm .
* Age ≥18 years.
* ECOG performance status ≤ 2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 6 weeks
* Participants must have normal organ and marrow function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

  * Adequate Organ Function Laboratory Values

    * Hematological

      ---- Absolute neutrophil count (ANC) ≥1,500 /mcL

      ---- Platelets ≥100,000 / mcL

      ---- Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
    * Renal

      ---- Serum creatinine ≤1.5 X upper limit of normal (ULN)

      ----- OR

      ---- Measured or calculated a creatinine clearance ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl)
    * Hepatic

      ---- Serum total bilirubin ≤ 1.5 X ULN

      ----- OR

      ---- Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN

      ---- AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN

      ----- OR

      ---- ≤ 5 X ULN for subjects with liver metastases
    * Albumin >2.5 mg/dL
    * Coagulation ---- International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

      * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
      * Creatinine clearance should be calculated per institutional standard.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document.
* Stable dose of dexamethasone 2mg or less for 7 days prior to initiation of treatment
* Patients may have progressive systemic disease
* Patients with untreated spinal cord metastases are eligible if lesions are asymptomatic
* Patients with untreated brainstem metastases are eligible if lesions are small and asymptomatic
* Cohort Specific Eligibility Criteria

  * Cohort A:

    * Measurable CNS disease (one parenchymal lesion ≥5 mm)
    * Previously untreated asymptomatic brain metastases
    * Patients with newly diagnosed, previously untreated primary tumors that present with brain metastases should not forego available therapy that has demonstrated a definitive overall survival benefit as firstline therapy for metastatic disease; therefore, in cases of previously untreated systemic solid tumors only those patients for whom there is no available therapy with definitive overall survival benefit, those that have failed at least one line of prior therapy for their primary tumor, or those refusing standard therapy will be eligible for this study. Specifically, for patients with previously untreated primary tumors, the following diagnoses will be excluded: HER2-positive breast cancer; small cell lung cancer; NSCLC with targetable genomic tumor aberrations (e.g. EGFR, ALK).
  * Cohort B:

    * Measurable CNS disease (one intracranial lesion ≥5 mm)
    * Progressive brain metastases after prior local CNS directed therapy such as radiation or surgery as defined by:

      * Untreated measurable lesions in patients that have received surgery and/or SRS to one or more other lesions
      * Residual or progressive lesions after surgery if asymptomatic
      * Patients who have had prior WBRT and/or SRS and then whose lesions have progressed are eligible. Lesions treated with SRS may be eligible if there is unequivocal evidence of progression
  * Cohort C:

    --- Carcinomatous meningitis, as defined by positive cytology
  * Cohort D:

    * Measurable CNS disease (one parenchymal lesion ≥5 mm)
    * 1-4 brain metastases (where stereotactic radiosurgery would be indicated)
    * Histologically confirmed diagnosis of melanoma

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days of protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Participants who are receiving any other investigational agents.
* Has a diagnosis of immunodeficiency.
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone >2mg/day or bioequivalent within 7 days of initiating therapy.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids as described in Section 3.2.4, within three months of start of study drug
* Hypersensitivity to pembrolizumab or any of its excipients
* Has a known history of active TB (Bacillus Tuberculosis)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Unable to undergo brain MRI.
* Participants who are receiving other concurrent chemotherapies or immunotherapies for their cancer (except for patients who will receive trastuzumab, bisphosphonates, denosumab or ovarian suppression therapy Radiation therapy to a symptomatic single metastatic site or to the brain may be allowed at the investigator's discretion).
* Will need immediate local surgery or radiation for their brain metastases
* Acute symptomatic CNS hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 Weeks
  Contrast-enhanced cranial MRI will be performed every 6 weeks. The proportion of patients in each cohort with a best response of CR or PR will be presented with a 90% confidence interval estimated using the method of Atkinson and Brown, which allows for the two-stage design.
Overall Survival Rate | 3 Months
  Any patient whose vital status is unknown due to loss of follow-up will be classified as having died for purposes of estimating the primary endpoint. The proportion of patients alive at six months will be summarized with a 90% confidence interval estimated using the method of Atkinson and Brown, which allows for the two-stage design.
Extracranial Overall Response Rate | 3 Months
  The proportion of patients with a best extracranial response of CR or PR will be presented with a 90% confidence interval estimated using the method of Atkinson and Brown, which allows for the two-stage design.

SECONDARY OUTCOMES:
Number of Participants with grade-3 or higher hematologic toxicities or grade-3 or higher neurologic toxicities | Baseline to 21 Days
Overall Survival Rate | 3 Months and 6 Months
  Kaplan-Meier
Intracranial Response Rate | 6 Months
  intracranial response (CR or PR by RANO) will be presented with a two-sided, 90% exact binomial confidence interval
Extracranial Response Rate | 6 Months
  Extracranial response rates (CR or PR) according to RECIST and irRC will be summarized for Cohorts A, B, C, and D
Extracranial PFS | 3 Months and 6 Months
Intracranial PFS | 3 Months and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Brastianos, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Priscilla Brastianos, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brastianos PK, Kim AE, Giobbie-Hurder A, Lee EQ, Lin NU, Overmoyer B, Wen PY, Nayak L, Cohen JV, Dietrich J, Eichler A, Heist RS, Krop I, Lawrence D, Ligibel J, Tolaney S, Mayer E, Winer E, Bent B, de Sauvage MA, Ijad N, Larson JM, Marion B, Nason S, Murthy N, Ratcliff S, Summers EJ, Mahar M, Shih HA, Oh K, Cahill DP, Gerstner ER, Sullivan RJ. Pembrolizumab in brain metastases of diverse histologies: phase 2 trial results. Nat Med. 2023 Jul;29(7):1728-1737. doi: 10.1038/s41591-023-02392-7. Epub 2023 Jun 2. PMID 37268724
- [Derived] Brastianos PK, Lee EQ, Cohen JV, Tolaney SM, Lin NU, Wang N, Chukwueke U, White MD, Nayyar N, Kim A, Alvarez-Breckenridge C, Krop I, Mahar MK, Bertalan MS, Shaw B, Mora JL, Goss N, Subramanian M, Nayak L, Dietrich J, Forst DA, Nahed BV, Batchelor TT, Shih HA, Gerstner ER, Moy B, Lawrence D, Giobbie-Hurder A, Carter SL, Oh K, Cahill DP, Sullivan RJ. Single-arm, open-label phase 2 trial of pembrolizumab in patients with leptomeningeal carcinomatosis. Nat Med. 2020 Aug;26(8):1280-1284. doi: 10.1038/s41591-020-0918-0. Epub 2020 Jun 2. PMID 32483359